CLINICAL TRIAL: NCT03011632
Title: The Role of Nonspecific Immune Response of the Airway Mucosa in Children With Chronic Rhinosinusitis and Asthma
Brief Title: Response of the Airway in Sinusitis and Asthma
Acronym: RAISe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Pawel Majak, MD, PhD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNN/153/16/KE
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sinusitis; Asthma
MeSH Terms: conditions — Sinusitis; Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mometasone nasal (Experimental): a group of children who will receive a nasal mometasone in an atomiser for three months (one application, once per day) and supplemental 3ml 0.9% sodium chloride (NaCl) solution in a nasal nebuliser once a day for 3 months,
  Interventions: Drug: Mometasone Nasal
- placebo mometasone (Placebo Comparator): a group of children without immunoglobulin E (IgE) - dependent hypersensitivity who will receive nasal mometasone placebo in an atomiser for three months (one application, once per day) and supplemental 3ml 0.9% NaCl solution in a nasal nebuliser once a day for 3 months,
  Interventions: Drug: placebo mometasone

INTERVENTIONS:
Drug: Mometasone Nasal — a group of children who will receive a nasal mometasone in an atomiser for three months (one application, once per day) and supplemental 3ml 0.9% Sodium chloride (NaCl) solution in a nasal nebuliser once a day for 3 months
  Other Names: NasometinTM, Sandoz
  Arms: mometasone nasal
Drug: placebo mometasone — a group of children without IgE-dependent hypersensitivity who will receive nasal mometasone placebo in an atomiser for three months (one application, once per day) and supplemental 3ml 0.9% NaCl solution in a nasal nebuliser once a day for 3 months,
  Other Names: placebo
  Arms: placebo mometasone

SUMMARY:
The project is intended to be realised in two phases. In the first stage, a case control study will be performed. In the second phase, double-blind, placebo controlled study will be conducted. In the first phase 3 groups of children will be compare: i) a group of children suffering from chronic rhinosinusitis (CRS) (fulfilling the European Position Paper on Rhinosinusitis and Nasal Polyps (EPOS) criteria) and asthma (fulfilling the Asthma Predictive Index (API) criteria) (CRS+/asthma+, n=90), ii) a group of children suffering from CRS (fulfilling the EPOS criteria) but without asthma symptoms (negative API criteria) (CRS+/asthma-, n=30) and iii) a group of children without symptoms of CRS (negative EPOS criteria) and without asthma symptoms (negative API criteria) (CRS-/asthma-, n=30). In the second phase the effect of intranasal glucocorticosteroids will be assessed. The following research methods will be used: CRS-symptom score questionnaire (SN-5) and Childhood Asthma Control Test (cACT) questionnaires, skin prick test, spirometry, measurement of nitric oxide NO in exhaled breath (FeNO), taste perception test, eosinophil morphology assessment, ratio: glucose concentration in nasal secretion/serum glucose level, concentration of specific immunoglobulin (Ig) E, total immunoglobulin G (IgG) and immunoglobulin A (IgA), the proportion of innate lymphoid cells (ILC) and regulatory lymphocytes cells in the peripheral blood. Endoscopic examination of the upper airways will be performed and samples of the mucosa will be taken. The mucosal examination will be as follows: i) polymerase chain reaction (PCR) examination for the detection of the presence of viral and bacterial genetic material, ii) measurement of the expression of the various messenger ribonucleic acid (mRNA), iii) measurement of the expression of mRNA for the Epithelial-Mesenchymal Transition (EMT) genes and iv) percentage of ILCs.

DETAILED DESCRIPTION:
Persistence of CRS and asthma require multiple interconnected feedback and feed-forward circuits between ILCs and epithelial cells. It seems that type 2 ILCs (ILC2) are the most important accelerators of type II immune response that prepare cytokine microenvironment for Th2 cells chronic activation. What decide on ILC2 accumulation - this is an urgent question. The aim of the proposed project is to examine the role of the innate immune response of airways in children suffering from chronic rhinosinusitis and asthma.

The project is intended to be realised in two phases. In the first stage, a case control study will be performed. In the second phase, double-blind, placebo controlled study will be conducted. In the first phase 3 groups of children will be compare: i) a group of children suffering from CRS (fulfilling the EPOS criteria) and asthma (fulfilling the API criteria) (CRS+/asthma+, n=90), ii) a group of children suffering from CRS (fulfilling the EPOS criteria) but without asthma symptoms (negative API criteria) (CRS+/asthma-, n=30) and iii) a group of children without symptoms of CRS (negative EPOS criteria) and without asthma symptoms (negative API criteria) (CRS-/asthma-, n=30). In the second phase the effect of intranasal glucocorticosteroids will be assessed. The following research methods will be used: SN-5 and cACT questionnaires, skin prick test, spirometry, measurement of NO in exhaled breath, taste perception test, eosinophil morphology assessment, ratio: glucose concentration in nasal secretion/serum glucose level, concentration of specific immunoglobulin E, total IgG and IgA, the proportion of ILC2 cells and regulatory cells in the peripheral blood. Endoscopic examination of the upper airways will be performed and samples of the mucosa will be taken. The mucosal examination will be as follows: i) PCR examination for the detection of the presence of viral and bacterial genetic material, ii) measurement of the expression of the various mRNA types, iii) measurement of the expression of mRNA for the Epithelial-Mesenchymal Transition (EMT) genes and iv) percentage of ILC 1, 2 and 3 cells and regulatory cells.

ELIGIBILITY:
Inclusion Criteria:

* a group of children (n=90) suffering from CRS (fulfilling the EPOS criteria, European Position Paper on Rhinosinusitis and Nasal Polyps) and asthma (fulfilling the API criteria, Asthma Predictive Index), including a 30-person subgroup diagnosed with clinically significant IgE-dependent hypersensitivity (accordance between symptoms and current exposure to sensitizing allergen),
* a group of children (n=30) suffering from CRS (fulfilling the EPOS criteria) but without asthma symptoms (negative API criteria), including a 15-person subgroup diagnosed with clinically significant IgE-dependent hypersensitivity (accordance between symptoms and current exposure to sensitizing allergen),
* a group of children (n=30) without symptoms of CRS (negative EPOS criteria) and without asthma symptoms (negative API criteria).

Exclusion Criteria:

* food allergy with symptoms affecting the respiratory tract
* contraindication to nasal endoscopy or contraindication to nasal mucosa biopsy
* hypertrophy of the third tonsil exceeding 60% of the nasopharynx (the criterion of obstruction being an indication for adenoidectomy). In these patients, the anatomical nasal obstruction may be the single cause of chronic inflammation in the airways, and hence verification of the hypotheses is impossible
* confirmed immunodeficiency
* exacerbation of asthma requiring systemic administration of glucocorticosteroids
* obesity, exposure to tobacco smoke
* other chronic illnesses and clinical conditions, which in the opinion of the researcher may influence the evaluation and the course of the study.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test for children (cACT™) | 12 months
  Childhood Asthma Control Test (cACT™), will be used, which has been recommended by the Global Initiative for Asthma (GINA) Report
SN-5 | 12 months
  validated questionnaire for the assessment for quality of life in children with CRS (5 symptom-cluster items covering the domains of sinus infection, nasal obstruction, allergy symptoms, emotional distress, and activity limitations)

SECONDARY OUTCOMES:
Spirometry | 12 months
  Respiratory function tests will be performed according to the American Thoracic Society (ATS) standards. The best result of three spirometric maneuvers will be selected for the analysis of obstructive disorders and the level of disease severity according to the standards of the Polish Society of Lung Diseases. The analysis will include FEV1% (A/N% - the percent of the measured to predicted value).
Nasal fraction of exhaled nitric oxide (nFeNO) Measurements | 12 months
  Measurements of nasal fraction of exhaled nitric oxide (nFeNO) will be performed using an electrochemical analyzer (ExpAir) according to the manufacturer's instructions. The detection limit ranged from 1 ppb to 6000 ppb.
Glucose concentration | 12 months
  Glucose concentration in serum and in nasal secretions will be assessed using glucose oxidase sticks (Roche, Lewes, East Sussex, U.K.). Nasal glucose concentration will analyzed in the context of blood glucose level using following ratio: nasal glucose level/blood glucose level.
Immunophenotyping | 12 months
  Mucosa - The nasal mucosa sample will be gently processed (mechanical dissociation, mild enzyme digestion) to produce a single cell suspension. It will be further fixed and stained with specific cocktail of fluorescent dye-stained antibody and then cell identification will be performed by flow cytometry. The relative count of all cell subsets will be determined. All procedures will be performed in buffers containing brefeldin and/or monesin to prevent dislocation of proteins of interest.
quantitative polymerase chain reaction (qPCR) | 12 months
  Total RNA will be isolated from mucosa samples and then reverse-transcribed with e.g. Thermo Scientific Maxima Reverse Transcriptase. qPCR reaction will be performed using house-designed primer sets. Relative expression of genes of interest (involved in innate response) will be analyzed against selected house-keeping gene transcripts.
  Manufacturer recommended procedure will be used to quantify Human Epithelial to Mesenchymal Transition gene panel and Multiplex Real-Time PCR for pathogen genes

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Majak, MD, PhD, Principal Investigator — Department of Internal Medicine, Asthma and Alergology, Barlicki Hospital,
Locations (1):
- Department of Internal Medicine, Asthma and Allergy, Barlicki University Hospital, Medical University of Lodz, Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latek M, Lacwik P, Molinska K, Blauz A, Lach J, Rychlik B, Strapagiel D, Majak J, Molinska J, Czech D, Seweryn M, Kuna P, Palczynski C, Majak P. Effect of an Intranasal Corticosteroid on Quality of Life and Local Microbiome in Young Children With Chronic Rhinosinusitis: A Randomized Clinical Trial. JAMA Pediatr. 2023 Apr 1;177(4):345-352. doi: 10.1001/jamapediatrics.2022.6172. PMID 36848113
- [Derived] Molinska K, Latek M, Rychlik B, Lach J, Strapagiel D, Majak J, Blazowski L, Jerzynska J, Kuna P, Majak P. House dust mite sensitization and frequent antibiotic courses may suppress remission of rhinosinusitis and asthma symptoms in young children. Allergy. 2022 Jan;77(1):301-304. doi: 10.1111/all.15085. Epub 2021 Sep 17. No abstract available. PMID 34510485
- [Derived] Majak P, Molinska K, Latek M, Rychlik B, Wachulec M, Blauz A, Budniok A, Gruchala M, Lach J, Sobalska-Kwapis M, Baranowska M, Krolikowska K, Strapagiel D, Majak J, Czech D, Palczynski C, Kuna P. Upper-airway dysbiosis related to frequent sweets consumption increases the risk of asthma in children with chronic rhinosinusitis. Pediatr Allergy Immunol. 2021 Apr;32(3):489-500. doi: 10.1111/pai.13417. Epub 2020 Dec 18. PMID 33222307